CLINICAL TRIAL: NCT01391858
Title: Effects of Oral Pregabalin Versus Placebo on Postoperative Pain and Morphine Consumption After Mastectomy
Brief Title: Postoperative Pain and Morphine Consumption After Mastectomy - Lyrica
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Babatunde Ogunnaike, MD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2004-0643; NCT00631891 (obsolete NCT alias); NCT02213445 (obsolete NCT alias)
Record Dates: First submitted 2011-06-27; First posted 2011-07-12 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Post-operative Pain
Keywords: Pregabalin; Postoperative pain; Mastectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pregabalin (Active Comparator): pregabalin (lyrica)
  Interventions: Drug: lyrica
- placebo (Placebo Comparator): placebo
  Interventions: Drug: lyrica

INTERVENTIONS:
Drug: lyrica — 150mg of pregabalin/placebo
  Other Names: pregabalin

SUMMARY:
This study will compare the effects of oral pregabalin with placebo on postoperative pain and morphine usage after mastectomy.

Pregabalin is an anticonvulsant agent approved by the United States Food and Drug Administration (FDA) for the treatment of neuropathic pain associated with post-herpetic neuralgia and diabetic neuropathy.

Women 18-70 years of age, undergoing unilateral modified mastectomy or lumpectomy with axillary node dissection will be recruited to participate in the study. Patients unable to cooperative, those that have known allergy to pregabalin or morphine and a history of drug or alcohol abuse, chronic pain, history of daily intake of analgesics or steroids, or impaired kidney function will all be excluded from the study. A pregnancy test will also be performed to exclude pregnant women from the study.

Oral pregabalin 300 mg (or placebo) will be administered to patients 1-2 hours before surgery followed by 150 mg 12 hours later. Thereafter, 150 mg of oral pregabalin (or placebo) will be administered twice daily until day 14. Whether a patient receives pregabalin or placebo will be decided based on a process similar to tossing a coin.

Patients will receive a standard general anesthetic for their operation and will receive intravenous patient-controlled analgesia (PCA) morphine for pain in the immediate postoperative period. Oral opioids will be administered after discontinuation of the PCA.

Subjects will be visited after the operation while in the hospital and intermittently for three months at the outpatient clinic after discharge from the hospital. Subjects will be asked to return remaining study drug/empty container when they are at the hospital for their 2 week follow up visit.

Potential adverse effects of pregabalin include dizziness, somnolence, peripheral edema, weight gain, headache, dry mouth, blurry vision, and ataxia. The incidence of these side effects occurring ranges variously between 1 and 25%. Investigators will closely monitor all patients for the occurrence of these side effects.

DETAILED DESCRIPTION:
TITLE: The Effects of Oral Pregabalin versus Placebo on Postoperative Pain and Morphine Consumption after Mastectomy

INVESTIGATOR: Babatunde O. Ogunnaike, MD. Department of Anesthesiology and Pain Management, University of Texas Southwestern Medical Center at Dallas, Texas

RATIONALE: In recent years, persistent pain after surgical procedures has been recognized as a major factor delaying recovery and return to normal daily living. Long-lasting pain has been reported after numerous surgical procedures including mastectomy. The prevalence of persistent post-mastectomy pain has been quoted to be anywhere from 40% to 80% and may substantially impact the life of patients treated for cancer (Smith et al. Pain 1999; 83: 91-5). Peripheral and central sensitization after tissue and nerve injury have been implicated in the development of more intractable pain that potentially can become chronic (Joshi & Ogunnaike, Anesthesiology Clin N Am 2005; 23: 21-36) Gabapentin, an anticonvulsant widely used for the treatment of chronic pain, has been shown to decrease neuropathic pain (Rice & Maton, Pain 2001; 94: 215-24) Dirks et al. (Anesthesiology 2002; 97: 560) reported that gabapentin 1200 mg prior to surgery reduced postoperative morphine requirements and movement-related pain after radical mastectomy. However, the immediate as well as long-term benefits of the drug were not evaluated in their study. Fassoulaki et al. (Anesth Analg 2002; 95: 985-91) also observed that pain at rest and movement pain were both reduced by gabapentin in the early postoperative period. Pregabalin is a new anticonvulsant agent recently approved by the FDA for the treatment of neuropathic pain associated with post-herpetic neuralgia (PHN) and diabetic peripheral neuropathy (DPN) [Gajraj NM. Pain Practice 2005; 5: 95-102]. This study is designed to evaluate the analgesic efficacy of pregabalin after mastectomy.

OBJECTIVES:

Primary: To evaluate the effects of pregabalin on postoperative opioid requirements and opioid-related side effects Secondary: To evaluate the effects of pregabalin on pain scores at 3 months after mastectomy.

INCLUSION CRITERIA:

1. Women 18-70 years of age
2. American Society of Anesthesiologists (ASA) physical status I to III
3. Undergoing unilateral modified radical mastectomy or lumpectomy with axillary node dissection

EXCLUSION CRITERIA:

1. Patients unable to cooperate
2. Allergy to pregabalin or morphine
3. History of drug or alcohol abuse
4. Chronic pain
5. Daily intake of analgesics or steroids
6. Impaired kidney function

OTHER THERAPY: IV-PCA morphine for rescue pain management in the immediate postoperative period and oral opioids after discontinuation of IV-PCA. Patients will be started on morphine PCA at a dose of 1 mg every 10 minutes for a maximum possible total dose of 6 mg per hour. This dose of morphine can be increased at the discretion of the treating physician. Transition to oral opioid hydrocodone/acetaminophen (5 mg/500 mg) will begin at 8 am on postoperative day 1 at a dose of 1 tablet every 4 hours as needed for pain. Total dose of morphine and the total number of tablets of hydrocodone/acetaminophen will be recorded immediately prior to discharge.

STUDY DESIGN: Phase III, randomized, double-blind, placebo-controlled study.

STUDY DRUG REGIMENS: Oral pregabalin 300mg (or placebo) will be administered to patients 1-2 hours before surgery followed by 150mg 12 hours later. Thereafter, 150mg of oral pregabalin (or placebo) will be administered twice daily until day 14.

DURATION OF STUDY: Patients will be followed for 3 months (90 days)

VISIT FREQUENCY: Patients will be visited daily while in hospital and followed daily postoperatively via telephone for 1 week and thereafter on postoperative days 14, 30, and 90 approximately. After discharge home, patients will be contacted by telephone to record pain assessments. The patient will be asked to return remaining study/drug empty container at the hospital when she comes in for her 2 week follow up visit with the surgery oncology clinic.

SAMPLE SIZE: Based on previous studies, a 30% reduction in opioid use is considered to be clinically relevant, with a type 1 error of 5% and a power of 90%, 40 patients will be required in each study group.

EFFICACY MEASURES:

1. Pain scores (VAS) and categorical
2. Morphine consumption (IV-PCA and oral opioid dosage)
3. Side effects rated using the symptom distress questionnaire, which includes measure of frequency, intensity, and bothersomeness evaluated on a four-point verbal scale (none, mild, moderate, severe).
4. Modified Brief Pain Inventory - short form (mBPI - sf)

PATIENT SAFETY PROCESS AND MONITORING:

Safety assessments would include monitoring of adverse events, the occurrence, nature, intensity, and relationship to the study drug. Clinical experience with a group-related drug (gabapentin) and results from clinical trials with pregabalin supports the notion that pregabalin is very well tolerated with minimal side effects including, headache, dizziness, somnolence, blurring of vision, weight gain, and peripheral edema. Patients would be specifically questioned about these side effects and any other unanticipated occurrences during clinic visits and over the telephone. Patients would be advised to avoid consumption of alcohol which may potentiate the sedative effects of pregabalin. Patients that may be on central nervous system depressants such as opiates or benzodiazepines would be informed that they may experience additive central nervous system (CNS) effects such as somnolence. Patient who may become pregnant will be advised to notify the investigators so that they may be removed from the study.

REPORTING ADVERSE EVENTS Definition An adverse event is any condition, which appears or worsens after participation in the study. All adverse events will be noted on the Adverse Reaction Case Report Form, whether or not it is felt to be related to the trial activities.

Severity

Whenever possible adverse events will be graded by a numerical score according to the defined Toxicity Grading Scale (NCI's Common Toxicity Criteria). Adverse events not included in the defined toxicity Grading Scale will be scored on the Adverse Reaction CRF according to their impact on the subject's ability to perform daily activities as follows:

Mild (causing no limitation of usual activities) Grade 1 Moderate (causing limitation of usual activities) Grade 2 Severe (causing inability to carry out usual activities) Grade 3

Serious Adverse Events

International Conference on Harmonisation (ICH) Guideline E6 defines a serious adverse event as those events which meet any of the following criteria:

* Fatal
* Immediately life-threatening
* Results in inpatient hospitalization or prolongation of existing hospitalization
* Results in persistent or significant disability/incapacity
* Results in a congenital anomaly/birth defect

Follow-up All adverse events will be followed up according to good medical practices.

Adverse Event Reporting All adverse experiences occurring during participation in the trial will be reported on the Adverse Reaction form in the subject's Clinical Research File (CRF) binder. The nature of each adverse event, date and time of onset, outcome, intensity and action taken will be established. Details of any corrective treatment will be recorded on the appropriate pages of the CRF binder.

Any adverse event that is serious and unexpected will be reported within two days to the Simmons Comprehensive Cancer Center Data and Safety Monitoring Committee, the UT Southwestern Institutional Review Board, the UTSW Medical Risk Management Office, and the Study Sponsor (DoD).

Institutional Review Board: 214-648-3060 UT Southwestern Medical Risk Management Office: 214-648-6905 SCCC DSMC: 214-648-1906

Data and Safety Monitoring Plan

This protocol falls under the purview of The Simmons Comprehensive Cancer Center (SCCC) Data and Safety Monitoring Committee (DSMC). Data and safety monitoring will be conducted as described in the SCCC Operations Manual which is available on request. Briefly, The data and safety monitoring plan at the University of Texas Southwestern Medical Center (UTSW) Simmons Comprehensive Cancer Center is designed to ensure that the safety and data quality for clinical trials involving patients with cancer or trials for cancer control, screening or prevention, meet the requirements of UTSW, the SCCC, the UTSW Institutional Review Board (IRB), the National Cancer Institute (NCI) as well as local, state and federal regulations. The Data and Safety Monitoring Committee (DSMC) is an independent committee appointed by the Director of the Cancer Center and is responsible for carrying out the data and safety monitoring plan. The plan mandates daily monitoring of all Severe Adverse Events (SAE) reported in conjunction with trials conducted through the SCCC Clinical Research Office. Accrual and adverse events (not serious) are reviewed quarterly. The DSMC has the authority to recommend suspension of closure of a trial for safety or performance issues.

ELIGIBILITY:
Inclusion Criteria:

1. Women, 18-70 years of age
2. ASA physical status I to III
3. Undergoing unilateral modified radical mastectomy or lumpectomy with axillary node dissection

Exclusion Criteria:

1. Patients unable to cooperate
2. Have known allergy to pregabalin or morphine
3. A history of drug or alcohol abuse
4. History of chronic pain
5. Daily intake of analgesics or steroids
6. Impaired kidney function

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-12; Primary Completion 2012-11 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babatunde Ogunnaike, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In recent years, surgical techniques have evolved from mastectomy with lymph node dissections to other forms of less invasive or nonsurgical techniques and these changes reduced the number of patients getting an axillary lymph node dissection (personal communication with the study-associated surgeon).
Pre-assignment Details: A total of 80 patients were consented. 7 patients did not show up for surgery. Of the 73 patients randomized, only 49 received intervention. The remaining 24 either had their surgery cancelled, withdrew their consent before intervention, or did not receive the loading dose in time to continue with the study.
Groups:
- Pregabalin: Pregabalin 300 mg 1-2 hrs. before the surgery and then 150 mg twice a day for 14 days
- Placebo: Placebo 1-2 hrs. before the surgery and then twice daily for 14 days
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 25 | 24
Completed | 23 | 24
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (9) | 47 (8) | 49 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: The Postoperative Opioid Requirement After Mastectomy
Description: IV Patient Controlled Analgesia (PCA) morphine for rescue pain management in the immediate postoperative period for an average of 24 hrs after mastectomy
Time Frame: Participants received PCA pump, an average of 24 hrs after mastectomy
Measure: Median (Inter-Quartile Range); unit: milligram (mg)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 23 | 24
milligram (mg) | 9 [2 to 29] | 7.5 [2.4 to 23]

2. Primary Outcome: Oral Opioids Consumption
Description: Oral opioids consumption after mastectomy until hospital discharge.
Time Frame: Participants were followed for the consumption of oral opioid for the duration of hospital stay, an average of 3 days after mastectomy
Measure: Median (Inter-Quartile Range); unit: milligram (mg)
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 23 | 24
milligram (mg) | 5 [0 to 20] | 10 [5 to 20]

3. Secondary Outcome: Pain Scores
Description: Visual Analog Pain Scores (VAS); 0 (no pain) to 10 (worst possible pain)
Time Frame: Participants' pain score was assessed on the first postoperative day after mastectomy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 4 [0 to 7] | 4 [0 to 8]

4. Secondary Outcome: Pain Scores
Description: Visual Analog Pain Scores (VAS); 0 (no pain) to 10 (worst possible pain)
Time Frame: Participants' pain score was assessed at hospital discharge, an average of 3 days after mastectomy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 4 [0 to 6] | 4 [0 to 7]

5. Secondary Outcome: Pain Scores
Description: Visual Analog Pain Scores (VAS); 0 (no pain) to 10 (worst possible pain)
Time Frame: Participants' pain score was assessed after discharge on the 7th day after mastectomy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 3 [0 to 5] | 3 [0 to 6]

6. Secondary Outcome: Pain Scores
Description: Visual Analog Pain Scores (VAS); 0 (no pain) to 10 (worst possible pain)
Time Frame: Participants' pain score was assessed after discharge on the 14th day after mastectomy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 3 [0 to 5] | 2 [0 to 8]

7. Secondary Outcome: Pain Scores
Description: Visual Analog Pain Scores (VAS); 0 (no pain) to 10 (worst possible pain)
Time Frame: Participants' pain score was assessed after discharge on the 30th day after mastectomy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 2 [0 to 5] | 2 [0 to 6]

8. Secondary Outcome: Pain Scores
Description: Visual Analog Pain Scores (VAS); 0 (no pain) to 10 (worst possible pain)
Time Frame: Participants' pain score was assessed after discharge on the 90th day after mastectomy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 1 [0 to 8] | 1 [0 to 5]

ADVERSE EVENTS:
Time Frame: 90 days after mastectomy
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin (N=23) | Placebo (N=24)
Surgical wound hematoma (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Desaturation in the operating room (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Desaturation in the operating room leading to premature termination of surgery.
Erythema and streaking of left breast skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wound debridement (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient was admitted to wound care of incision site from left radical mastectomy. Surgery was performed debridement of the necrotic tissue.
Micrometastases to axilla (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Micrometastases to the right axilla, status post-mastectomy for infiltrating ductal carcinoma. Evaluated as not related to study drug.
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Anemia secondary to postoperative hemorrhage. Required re-exploration of right axilla and ligation of bleeding branch of thoracodorsal artery.
Nerve injury (Surgical and medical procedures) | 0 (0) | 1 (1) — Injury of thoracic nerve during surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes